CLINICAL TRIAL: NCT05434455
Title: Effects of Remote Ischemic Preconditioning(RIPC) on the Prevention of Postoperative Delirium in Patients Undergoing Cardiac Surgery: A Pilot Randomized Clinical Trial
Brief Title: Effect of RIPC on the Prevention of POD in Patients Undergoing Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2022RIPC-delirium
Record Dates: First submitted 2022-06-22; First posted 2022-06-28 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Postoperative Delirium; Cardiac Surgery
MeSH Terms: conditions — Emergence Delirium | interventions — Reperfusion

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIPC (Experimental): RIPC was induced with 3 cycles of 5 minutes of ischaemia and 5 minutes of reperfusion on the upper arm. By using blood pressure cuff inflation, patients in the RIPC group were exposed to a pressure 50 mmHg higher than the systolic radial artery pressure baseline.
  Interventions: Device: RIPC induced with 3 cycles of 5 minutes of ischaemia and 5 minutes of reperfusion
- Con (No Intervention): The control group had a deflated cuff placed on the upper arm for the same time.

INTERVENTIONS:
Device: RIPC induced with 3 cycles of 5 minutes of ischaemia and 5 minutes of reperfusion — RIPC was induced with 3 cycles of 5 minutes of ischaemia and 5 minutes of reperfusion on the upper arm. By using blood pressure cuff inflation, patients in the RIPC group were exposed to a pressure 50 mmHg higher than the systolic radial artery pressure baseline.
  Arms: RIPC

SUMMARY:
Postoperative delirium (POD) is one of the most frequent neurological complications in elderly patients and is closely associated with longer ICU stay and hospitalization, deterioration of long-term neurocognitive function, and increased mortality. The incidence of POD is significantly higher in elderly patients undergoing cardiac surgery than in other populations. Therefore, the prevention of POD is an important clinical problem to be solved urgently. In this study, we intend to observe the effect of RIPC on the prevention and treatment of POD in patients undergoing cardiac surgery through a prospective randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective cardiac surgery;
* age ≥ 18 yr;
* any sex;
* American Society of Anesthesiologists (ASA) class ≥II class;
* New York Heart Association (NYHA) ≥II class.

Exclusion Criteria:

* emergency surgery;
* a history of cardiovascular surgery;
* peripheral vascular disease affecting the upper limbs;
* acute myocardial infarction (MI) up to 14 days before surgery;
* a history of severe injuries and operations within 3 months before cardiac surgery;
* a history of cancer and chronic autoimmune diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-07-14 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | 7 days postoperatively or before discharge, whichever came first
  Patients were assessed for postoperative delirium by the Confusion Assessment Method (CAM) from the time they were transferred to the ICU at the end of surgery until 7 days postoperatively or before discharge, whichever came first

IPD SHARING:
Plan to Share IPD: Undecided